CLINICAL TRIAL: NCT03391570
Title: A Prospective Randomized Clinical Trial for Comparing Postoperative Pain Following COX-2 and Prostanoids Expression in Women Who Underwent Laparoscopic Surgery for Female Genital Disease
Brief Title: Comparing Postoperative Pain Following COX-2 and Prostanoids Expression
Acronym: COX2RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1477
Record Dates: First submitted 2017-10-24; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Female Genital Disease
Keywords: Laparoscopic surgery; COX-2 inhibitor; Celecoxib; Prostanoid
MeSH Terms: conditions — Genital Diseases, Female | interventions — Cyclooxygenase 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COX-2 inhibitor (Celecoxib) (Active Comparator): Celebrex; COX-2 inhibitor
  Interventions: Drug: COX-2 inhibitor; Procedure: Preoperative peritoneal biopsy; Procedure: Single-port laparoscopic surgery; Procedure: Postoperative peritoneal biopsy
- Placebo drug (Ramnos) (Placebo Comparator): Ramnos; Lactobacillus casei variety rhamnosus
  Interventions: Drug: Placebo Oral Tablet; Procedure: Preoperative peritoneal biopsy; Procedure: Single-port laparoscopic surgery; Procedure: Postoperative peritoneal biopsy

INTERVENTIONS:
Drug: COX-2 inhibitor — Celebrex 200mg/1cap 2 tablets, take medication an hour before surgery
  Arms: COX-2 inhibitor (Celecoxib)
Drug: Placebo Oral Tablet — Ramnos 250mg/1cap 2 tablets, take medication an hour before surgery
  Arms: Placebo drug (Ramnos)
Procedure: Preoperative peritoneal biopsy — Preoperative peritoneal biopsy (1x1cm sized peritoneal tissue)
Procedure: Single-port laparoscopic surgery — Single-port laparoscopic surgery with CO2 gas
Procedure: Postoperative peritoneal biopsy — Postoperative peritoneal biopsy (1x1cm sized peritoneal tissue)

SUMMARY:
The purpose of this study is to compare postoperative pain following COX-2 and prostanoids expression in women who underwent laparoscopic surgery for female genital disease in order to evaluate the effect of COX-2 on local inflammation, COX-2 and prostanoids expression followed by exposure time to carbon dioxide(CO2) gas, and degree of postoperative pain.

DETAILED DESCRIPTION:
In women who underwent laparoscopic surgery for female genital disease, the effect of COX-2 on local inflammation was assessed by randomization, using the COX-2 inhibitor celecoxib and placebo, comparative evaluation of expression of COX-2 and prostanoids by pre/postoperative peritoneal biopsy and postoperative pain depending on gas exposure time

ELIGIBILITY:
Inclusion Criteria:

* Female, Age ≥ 20 years
* Patients with benign female genital disease who need laparoscopic surgery
* Patients with benign disease who can be treated by single port laparoscopy
* Patients who signed an approved informed consent

Exclusion Criteria:

* Female, Age < 20 years
* Pregnancy
* Previous cancer history
* Patients who refuse to sign an informed consent
* Patients with benign female genital disease combined clinical peritonitis (ex. tubo-ovarian abscess, tubo-ovaritis, ruptured endometriosis)
* Patients with malignant female genital disease
* Patients who got surgery with multi-port laparoscopy
* Patients who are contraindicated with COX-2 inhibitors (liver disease, renal disease, active peptic ulcer, active gastrointestinal tract bleeding, ischemic heart disease, hyperkalemia)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change of biomarkers expression according to exposure to CO2 gas | Peritoneal biopsy will be done twice (intraoperative, at right after trocar insertion and right before trocar removal, an average of 2-3hours)
  Peritoneal biopsy and real-time polymerase chain reaction(RT-PCR), Immunohistochemistry of Biomarkers (COX-2, PGE2, PGF2, PGI2, TXA2)

SECONDARY OUTCOMES:
Visual analogue scale(VAS) score | every six hours for 48 hours
  Degree of postoperative pain (No pain : 0 / Moderate pain : 5 / Unbearable pain : 10)
Numbers of rescue analgesia | From postoperation state to discharge (up to 2 days)
  Frequency of additional pain killer (Tramadol 50mg, Ketorolac 2mg/kg)
Postoperative complication | From postoperation state to discharge (up to 2 days)
  nausea, vomiting, etc.
Duration of hospitalization | From postoperation state to discharge (up to 2 days)
  duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han KH, Park S, Lee S, Ham J, Lim W, Song G, Kim HS. Upregulation of 15-Hydroxyprostaglandin Dehydrogenase by Celecoxib to Reduce Pain After Laparoendoscopic Single-Site Surgery (POPCORN Trial): A Randomized Controlled Trial. Biomedicines. 2025 Jul 21;13(7):1784. doi: 10.3390/biomedicines13071784. PMID 40722854